CLINICAL TRIAL: NCT02392702
Title: A Two-Part Open-Label, Randomized, Sequential, Crossover, Single Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of C-10355 and C-10358 in Healthy Volunteers, With a PK Comparison to Kalydeco®
Brief Title: Study to Evaluate Safety, Tolerability and PK of C-10355 and C-10358 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Concert Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CP656.1001
Record Dates: First submitted 2015-03-05; First posted 2015-03-19 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Healthy
Keywords: Subjects; Safety/Efficacy Study; Randomized; Open Label
MeSH Terms: interventions — ivacaftor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- C-10355, 25 mg (Active Comparator): single oral dose.
  Interventions: Drug: C-10355
- C-10358, 25 mg (Active Comparator): single oral dose.
  Interventions: Drug: C-10358
- C-10355 or C-10358, 75 mg (Active Comparator): single oral dose.
  Interventions: Drug: C-10355; Drug: C-10358
- C-10355 or C-10358, 150 mg (Active Comparator): single oral dose.
  Interventions: Drug: C-10355; Drug: C-10358
- Kalydeco, 150 mg (Active Comparator): single oral dose.
  Interventions: Drug: Kalydeco
- C-10355 or C-10358, 300 mg (Active Comparator): single oral dose.
  Interventions: Drug: C-10355; Drug: C-10358

INTERVENTIONS:
Drug: C-10355
  Arms: C-10355 or C-10358, 150 mg; C-10355 or C-10358, 300 mg; C-10355 or C-10358, 75 mg; C-10355, 25 mg
Drug: C-10358
  Arms: C-10355 or C-10358, 150 mg; C-10355 or C-10358, 300 mg; C-10355 or C-10358, 75 mg; C-10358, 25 mg
Drug: Kalydeco
  Arms: Kalydeco, 150 mg

SUMMARY:
This two-part study will assess, in healthy volunteers, under both fasted and fed conditions, and in a sequential manner, the safety, tolerability and pharmacokinetics (PK) profile of single doses of C-10355 and C-10358 and single ascending doses of the selected compound compared to a single dose of Kalydeco®.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults between 18 and 50 years of age, inclusive
* Body weight ≥ 50 kg and BMI within the range of 18 to 30 kg/m2, inclusive, at screening

Exclusion Criteria:

* History of clinically significant central nervous system (eg, seizures), cardiac, pulmonary, metabolic, renal (including nephrolithiasis), hepatic, including history of Gilbert's syndrome or gastrointestinal (GI) conditions
* PR interval ≥ 220 msec or QRS duration ≥ 120 msec or QTcF interval > 450 msec obtained at screening visit or prior to the first dose of study drug
* Liver function tests greater than the upper limit of normal.
* Positive blood screen for human immunodeficiency virus (HIV antibody), hepatitis B virus surface antigen, or hepatitis C virus antibody at screening
* Urinalysis positive for greater than trace blood, protein or glucose
* A positive screen for alcohol, drugs of abuse, or tobacco use.
* Inability to comply with food and beverage restrictions during study participation.
* Donation or blood collection or acute loss of blood prior to screening.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2015-03; Primary Completion 2015-06 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 24 hours
  adverse events categorized by body system and MedDRA term
Pharmacokinetic Profile | 96 hours
  Measure exposure of test articles using area under the concentration time curve (AUC), maximum concentration (Cmax), half life (T 1/2)

CONTACTS AND LOCATIONS:
Overall Officials: Lana Pilja, Study Director — Concert Pharmaceuticals, Inc.
Locations (1):
- CMAX, Adelaide, South Australia, Australia